CLINICAL TRIAL: NCT06864377
Title: Ventral Hernia Improvement of Treatment and Life
Acronym: VITAL
Status: Enrolling by invitation | Type: Observational
Sponsor: Line Marker (Other)
Collaborators: Aage og Johanne Louis-Hansens Fond (Other)
Responsible Party: Sponsor-Investigator, Line Marker, Principal Investigator, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Other Study IDs: p-2024-17652
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Incisional Hernia; Parastomal Hernia; Ventral Hernia
Keywords: Incisional hernia; Parastomal hernia; Quality of life; Patient-reported outcomes
MeSH Terms: conditions — Incisional Hernia; Hernia, Ventral | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with incisinal hernias: Patients with incisional hernias who are either offered surgery or conservative treatment
- Patients with parastomal hernias: Patients with parastomal hernias who are either offered surgery or conservative treatment

INTERVENTIONS:
Other: Quality of life questionnair — The questionnaire used is the Abdominal Hernia Q, which is specific to ventral hernias. Patients will receive the questionnaire at baseline and at 1, 3, 6, and 12 months after ventral hernia repair. If treated conservatively, the questionnaire will be administered at 1, 3, 6, and 12 months after completing the baseline questionnaire.
  Other Names: Patient reported outcome

SUMMARY:
The goal of this clinical trial called the VITAL study is to learn if surgery has a positive impact on the quality of life in patients with incisional or parastomal hernia. The main questions it aims to answer are:

Does surgery alleviate patients from their initial problem? Does new discomfort arise after surgery? Do the symptoms worsen, and does quality of life deteriorate in patients who are not offered surgery? The project will also look at time to surgery and postoperative complications. Researchers will send questionnaires to the patients to answer.

Participants will:

Answer the baseline questionnaire. Answer the follow-up questionnaires at 1 month, 3 months, 6 months, 1 year, and 3 years after surgery or after the baseline questionnaire has been completed for those patients being managed conservatively with observation

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Incisional hernia or parastomal hernia

Exclusion Criteria:

- Can't understand or read Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred with a ventral hernia to the surgical outpatient clinic at Zealand University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life after ventral hernia repair for pateints with incisional hernia | From enrollment to the end of follow-up at 36 months.
  The patients will receive a questionnaire at baseline and at 1, 3, 6, 12, and 36 months of follow-up. The project will use the Abdominal Hernia-Q. It features both a pre- and postoperative form, including a total of 24 items with responses scored on a 4-point Likert scale. Patient responses will be averaged, producing a possible score range of 0 to 4.
Quality of life in patient with incisional hernia | From enrollment to the end of follow-up at 36 months.
  The patients will receive a questionnaire at baseline and at 1, 3, 6, 12, and 36 months of follow-up. The project will use the Abdominal Hernia-Q. It features both a pre- and postoperative form, including a total of 24 items with responses scored on a 4-point Likert scale. Patient responses will be averaged, producing a possible score range of 0 to 4.
Quality of life in patients with parastomal hernia | From enrollment to the end of follow-up at 36 months.
  The patients will receive a questionnaire at baseline and at 1, 3, 6, 12, and 36 months of follow-up. The project will use the Abdominal Hernia-Q. It features both a pre- and postoperative form, including a total of 24 items with responses scored on a 4-point Likert scale. Patient responses will be averaged, producing a possible score range of 0 to 4.
Changes in quality of life after ventral hernia repair in patients with parastomal hernia | From enrollment to the end of follow-up at 36 months.
  The patients will receive a questionnaire at baseline and at 1, 3, 6, 12, and 36 months of follow-up. The project will use the Abdominal Hernia-Q. It features both a pre- and postoperative form, including a total of 24 items with responses scored on a 4-point Likert scale. Patient responses will be averaged, producing a possible score range of 0 to 4.

SECONDARY OUTCOMES:
Time to surgery | From enrollment to the end of follow-up at 36 months.
  Days or months from the indication of surgery being set to ventral hernia repair.
Postoperative complications | From enrolment to the end of follow-up at 36 months
  Any adverse events or conditions that occur following a surgical procedure.
Risk of emergency surgery during the waiting time | From enrollment to the end of follow-up at 36 months
  Number of patients who are undergoing emergency surgery during the waiting time for planned surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, DMSc, Study Director — Zealand University Hospital, Køge; Line Marker, MD, Principal Investigator — Zealand University Hospital, Køge; Pernille D.K. Diasso, MD, Ph.d., Study Director — Zealand University Hospital, Køge
Locations (1):
- Department of surgery, Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following the review and approval of a research proposal and Statistical Analysis Plan (SAP), along with the execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Liang MK, Holihan JL, Itani K, Alawadi ZM, Gonzalez JR, Askenasy EP, Ballecer C, Chong HS, Goldblatt MI, Greenberg JA, Harvin JA, Keith JN, Martindale RG, Orenstein S, Richmond B, Roth JS, Szotek P, Towfigh S, Tsuda S, Vaziri K, Berger DH. Ventral Hernia Management: Expert Consensus Guided by Systematic Review. Ann Surg. 2017 Jan;265(1):80-89. doi: 10.1097/SLA.0000000000001701. PMID 28009730
- [Background] Pernar LIM, Pernar CH, Dieffenbach BV, Brooks DC, Smink DS, Tavakkoli A. What is the BMI threshold for open ventral hernia repair? Surg Endosc. 2017 Mar;31(3):1311-1317. doi: 10.1007/s00464-016-5113-5. Epub 2016 Jul 20. PMID 27440197
- [Background] Huntington C, Gamble J, Blair L, Cox T, Prasad T, Lincourt A, Augenstein V, Heniford BT. Quantification of the Effect of Diabetes Mellitus on Ventral Hernia Repair: Results from Two National Registries. Am Surg. 2016 Aug;82(8):661-71. PMID 27657579
- [Background] Borad NP, Merchant AM. The effect of smoking on surgical outcomes in ventral hernia repair: a propensity score matched analysis of the National Surgical Quality Improvement Program data. Hernia. 2017 Dec;21(6):855-867. doi: 10.1007/s10029-017-1664-1. Epub 2017 Sep 1. PMID 28864961
- [Background] Parker SG, Mallett S, Quinn L, Wood CPJ, Boulton RW, Jamshaid S, Erotocritou M, Gowda S, Collier W, Plumb AAO, Windsor ACJ, Archer L, Halligan S. Identifying predictors of ventral hernia recurrence: systematic review and meta-analysis. BJS Open. 2021 Mar 5;5(2):zraa071. doi: 10.1093/bjsopen/zraa071. PMID 33839749
- [Background] Henriksen NA, Bisgaard T, Andersen HF, Jorgensen LN, Helgstrand F. [Surgical treatment algorithm for ventral hernias]. Ugeskr Laeger. 2018 Sep 10;180(37):V02180096. Danish. PMID 30259832
- [Background] Sando A, Rosen MJ, Heniford BT, Bisgaard T. Long-term patient-reported outcomes and quality of the evidence in ventral hernia mesh repair: a systematic review. Hernia. 2020 Aug;24(4):695-705. doi: 10.1007/s10029-020-02154-1. Epub 2020 Mar 9. PMID 32152807
- [Background] Mohamud AA, Sando A, Helgstrand F, Bisgaard T. [Patient-reported outcome measures after ventral hernia surgery]. Ugeskr Laeger. 2021 Jan 4;183(1):V05200399. Danish. PMID 33491623
- [Background] Friis-Andersen H, Bisgaard T. The Danish Inguinal Hernia database. Clin Epidemiol. 2016 Oct 25;8:521-524. doi: 10.2147/CLEP.S99512. eCollection 2016. PMID 27822094
- [Background] Bisgaard T, Helgstrand F, Friis-Andersen H, Rosenberg J, Jørgensen LN, Pedersen KF, m.fl. Optimizing outcomes after hernia repair: scientific highlights from the Danish Hernia Database 2010-2020. Laparosc Surg. januar 2022;6:5-5.
- [Background] Helgstrand F, Jorgensen LN. The Danish Ventral Hernia Database - a valuable tool for quality assessment and research. Clin Epidemiol. 2016 Oct 25;8:719-723. doi: 10.2147/CLEP.S99501. eCollection 2016. PMID 27822119
- [Background] Bisgaard T, Kehlet H, Bay-Nielsen MB, Iversen MG, Wara P, Rosenberg J, Friis-Andersen HF, Jorgensen LN. Nationwide study of early outcomes after incisional hernia repair. Br J Surg. 2009 Dec;96(12):1452-7. doi: 10.1002/bjs.6728. PMID 19918863
- [Background] Kokotovic D, Bisgaard T, Helgstrand F. Long-term Recurrence and Complications Associated With Elective Incisional Hernia Repair. JAMA. 2016 Oct 18;316(15):1575-1582. doi: 10.1001/jama.2016.15217. PMID 27750295
- [Background] Manole TE, Daniel I, Alexandra B, Dan PN, Andronic O. Risk Factors for the Development of Parastomal Hernia: A Narrative Review. Saudi J Med Med Sci. 2023 Jul-Sep;11(3):187-192. doi: 10.4103/sjmms.sjmms_235_22. Epub 2023 Jul 15. PMID 37533654
- [Background] Deerenberg EB, Henriksen NA, Antoniou GA, Antoniou SA, Bramer WM, Fischer JP, Fortelny RH, Gok H, Harris HW, Hope W, Horne CM, Jensen TK, Kockerling F, Kretschmer A, Lopez-Cano M, Malcher F, Shao JM, Slieker JC, de Smet GHJ, Stabilini C, Torkington J, Muysoms FE. Updated guideline for closure of abdominal wall incisions from the European and American Hernia Societies. Br J Surg. 2022 Nov 22;109(12):1239-1250. doi: 10.1093/bjs/znac302. PMID 36026550
- [Background] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861
- See also: Annual Report 2023 from the Danish Hernia database — https://www.herniedatabasen.dk/_files/ugd/02befe_537096ef6bb64c56afa93214cbb0e77d.pdf